CLINICAL TRIAL: NCT01292018
Title: A Non Interventional, Cross Sectional, Epidemiological Study on the Management of Dyslipidemia in Type 2 DM Adult Patients in India
Brief Title: Management of Dyslipidemia in Adult Type 2 Diabetes Patients in India
Acronym: SOLID
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CIN-DUM-2010/1
Record Dates: First submitted 2011-01-31; First posted 2011-02-09 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Dyslipidemia; Type 2 Diabetes Mellitus
Keywords: Management of dyslipidemia in Type 2 Diabetes Mellitus adult patients in India; Dyslipidemia control rates in Type 2 diabetic Mellitus patients
MeSH Terms: conditions — Dyslipidemias; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Lipid profile ( Low Density Lipoproteins(LDL), High Density Lipoprotein (HDL), Triglycerides & Total cholesterol) Blood Glucose Measurements (Fasting Plasma Glucose)
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of study to assess the control of dyslipidemia in the Indian diabetic population treated with any hypolipidemic agent.

ELIGIBILITY:
Inclusion Criteria:

* Adult who is a known Type 2 diabetic as per the ADA 2010 criteria OR controlled diabetic (taking any antidiabetic medication)
* Patients in the study will have been on lipid lowering drugs at a stable dose for the last three months before the designated study visit.

Exclusion Criteria:

* Type 1 diabetic patients
* Patients with a history of hepatic or renal diseases
* Hypertension due to organic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 Diabetics with dyslipidemia on stable dose of Lipid Lowering Drugs(LLDs).
Sampling Method: Non-Probability Sample
Enrollment: 5400 (Actual)
Dates: Start 2011-02; Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Proportion of type 2 diabetic dyslipidemia patients achieving the target LDL goal according to ADA 2010. These patients should be on stable dose of Lipid Lowering Drugs(LDL) for at least 3 months

SECONDARY OUTCOMES:
Proportion of dyslipidemia control rate according to american diabetes Association (ADA) 2010 criteria by age and gender
Control of dyslipidemia by Lipid Lowering Drugs (LLDs) drugs alone or combination
Control of dyslipidemia by all commercial available brands hypolipidemics drugs